CLINICAL TRIAL: NCT03767283
Title: Genetic Characterization of Plasmids Carrying Carbapenemases and Quinolone Resistance Determinants in Klebsiella Pneumoniae Isolates in Assiut University Hospitals
Brief Title: Carbapenem and Quinolone Resistance in Klebsiella Pneumoniae
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Ali Ahmed, principle investigator, Assiut University
Other Study IDs: HAA
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Antibiotic Resistant Strain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Klebsiella pneumoniae is an important pathogen that frequently causes nosocomial community-acquired and infections, including pneumonia, urinary tract infections, bloodstream infections, pyogenic liver abscesses, and septic shock.

An emerging co-existence of carbapenems and fluoroquinolone resistance in Klebsiella pneumoniae is causing major difficulty in treating infections caused by such pathogen

DETAILED DESCRIPTION:
Plasmid mediated carbapenem resistance is mainly due to production of carbapenemase which belong to three classes of β-lactamases, the Ambler class A, B and D β -lactamases, among which the New Delhi metallo-β -lactamase has attracted significant attention in the last five years. New Delhi metallo-β -lactamase-1 is a class B metallo-β-lactamase and was first identified from a Klebsiella pneumoniae strain in 2008.

New Delhi metallo-β -lactamase-1 is frequently associated with other resistance genes, such as extended spectrum β- lactamase genes and plasmid-mediated quinolone resistance genes, which allows bacteria to gain resistance to different classes of antimicrobial agents simultaneously.

Plasmids and Integrons are mobile genetic elements that carry antimicrobial resistance genes. Horizontal transfer of those mobile genetic elements has been considered as one of the most important mechanisms for the dissemination of multi-drug resistance among bacteria.

Classification of plasmids on the basis of molecular typing and phylogenetic relatedness may help understand the distribution of plasmid types, the relationships involving plasmids carrying antimicrobial resistance genes. Plasmids can be classified into incompatibility groups by replicon typing or into types (clusters) by restriction fragment length polymorphism analysis.

Integrons act as genetic platform, which allow capture and expression of antibiotic resistance genes. There are 3 classes of integrons that are responsible for multi-drug resistance, which are classified based on the sequence of the integrase gene. Class 1 integrons are the most widespread class in Gram-negative bacteria.

One approach to preventing multi drug resistant infections is combination of two or more antimicrobial drugs during a treatment regimen . The combination of imipenem plus ciprofloxacin had shown Synergistic effect .

Loading of antibacterial agents into nanoparticles is one of the most promising approaches to reduce anti-microbial resistance. Nano formulations could enhance the intracellular bioavailability of the antimicrobial drugs, and, thus, decreasing the development of resistance. Moreover, the potential antibacterial activity of some nanoparticle-forming polymers might further increase the potency of the antibacterial drugs .

ELIGIBILITY:
Inclusion Criteria:

* admitted to intensive care unite

Exclusion Criteria:

* healthy

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with infections admitted to ICUs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-12-07 (Estimated)

PRIMARY OUTCOMES:
effect of combined antibiotic therapy on resistance | 1 year
  determination of minimum inhibitory concentration to antibiotics before and after combination

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Al-Marzooq F, Mohd Yusof MY, Tay ST. Molecular Analysis of Antibiotic Resistance Determinants and Plasmids in Malaysian Isolates of Multidrug Resistant Klebsiella pneumoniae. PLoS One. 2015 Jul 23;10(7):e0133654. doi: 10.1371/journal.pone.0133654. eCollection 2015. PMID 26203651
- [Background] Chang CY, Lin HJ, Chang LL, Ma L, Siu LK, Tung YC, Lu PL. Characterization of Extended-Spectrum beta-Lactamase-Carrying Plasmids in Clinical Isolates of Klebsiella pneumoniae from Taiwan. Microb Drug Resist. 2017 Jan;23(1):98-106. doi: 10.1089/mdr.2015.0212. Epub 2016 May 5. PMID 27148814
- [Background] Worthington RJ, Melander C. Combination approaches to combat multidrug-resistant bacteria. Trends Biotechnol. 2013 Mar;31(3):177-84. doi: 10.1016/j.tibtech.2012.12.006. Epub 2013 Jan 18. PMID 23333434
- [Background] Zhao JY, Zhu YQ, Li YN, Mu XD, You LP, Xu C, Qin P, Ma JL. Coexistence of SFO-1 and NDM-1 beta-lactamase genes and fosfomycin resistance gene fosA3 in an Escherichia coli clinical isolate. FEMS Microbiol Lett. 2015 Jan;362(1):1-7. doi: 10.1093/femsle/fnu018. Epub 2014 Dec 4. PMID 25790496